CLINICAL TRIAL: NCT06184516
Title: Assessment of Decision Tool to Select Women for Gynecologic Sparing Radical Cystectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-GU-008; OCR44653 (Other: University of Florida); IRB202400006 (Other: University of Florida)
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Carcinoma Bladder
Keywords: urothelial carcinoma; radical cystectomy; organ preservation; female
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reproductive organ sparing radical cystectomy (Experimental)
  Interventions: Procedure: Reproductive organ sparing radical cystectomy
- Radical cystectomy (Active Comparator)
  Interventions: Procedure: Radical cystectomy

INTERVENTIONS:
Procedure: Reproductive organ sparing radical cystectomy — Participants on this arm will undergo a reproductive organ sparing radical cystectomy if they are classified as "favorable" based on the decision tool.
  Arms: Reproductive organ sparing radical cystectomy
Procedure: Radical cystectomy — Participants on this arm will undergo a radical cystectomy if they are classified as "unfavorable" based on the decision tool.
  Arms: Radical cystectomy

SUMMARY:
Currently, the standard of care for female patients undergoing radical cystectomy includes the removal of the bladder, pelvic lymph nodes, anterior vagina, uterus, fallopian tubes and ovaries. Removal of female ancillary organs, both in pre and post-menopausal stages is associated with reduction in various quality of life metrics, including sexual health, cognitive decline and depression. Furthermore, removal of ovaries has been associated with increased cardiovascular events, metabolic acidosis, osteoporosis and bone fractures. In premenopausal women, the removal of the ovaries is associated with increased all-cause mortality. From an oncologic standpoint, multi institutional retrospective reviews have demonstrated certain pre-operative radiographic and cystoscopic risk factors that are associated with bladder cancer involvement of female reproductive organs. The absence of these unfavorable risk factors may provide an opportunity to spare women from undergoing unnecessary reproductive organ removal during RC. In doing so, this may eliminate the associated sequelae of removing these additional organs while also providing acceptable oncologic care. The investigators thus propose a decision tool to stratify women undergoing radical cystectomy as favorable and unfavorable for reproductive organ sparing radical cystectomy. This decision tool classification will be used to decide which patients will undergo reproductive organ sparing radical cystectomy versus radical cystectomy in this study.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ eighteen years of age
* Histologically proven diagnosis of urothelial carcinoma of the bladder, including variant histology
* Surgical candidate for radical cystectomy
* Be able to undergo pelvic MRI. Minimum standards for MRI imaging will include the following:

  * MRI of the pelvis on 1.5T or higher strength magnet.
  * T2 weighted imaging in multiple planes.
  * T1 weighted imaging pre and post contrast administration (unless contrast is contraindicated by allergy or renal insufficiency)
* Cystoscopic evaluation completed by urologist within 120 days prior to surgery (ROS-RC or RC)
* Staging imaging within 90 days prior to surgery (ROS-RC or RC). If receiving neoadjuvant therapy prior to surgery (ROS-RC or RC), repeat staging imaging must be completed after the neoadjuvant therapy is completed, or no longer tolerated by the patient.
* Staging imaging must include MRI of the pelvis within 90 days of surgery (ROS-RC or RC)
* Written informed consent obtained from the subject and the ability for the subject to comply with all the study-related procedures.
* Presence of at least one or more ancillary organs. Ancillary organs defined as anterior vagina, uterus, fallopian tubes (only 1 tube present will be considered at physician discretion), and ovaries.
* ECOG Performance Status of 0-2

Exclusion Criteria:

* Patients with regional or distant metastatic disease
* Non-urothelial bladder cancer.
* Not a surgical candidate for radical cystectomy
* Unable to have MRI of pelvis that meets the minimum standards in the inclusion criteria above.
* Subjects of childbearing potential (SOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy during study intervention and for at least 12 weeks after the study intervention.
* Patients with other known active malignancies which may confound the recurrence rates
* Patients with known germline mutations in DNA damage repair genes (BRCA1/BRCA 2)
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.
* Subjects who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for complications, in the opinion of the treating physician.
* Administration of a vaccine containing live virus within 30 days prior to the study intervention. Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose. Non-live versions of the COVID vaccine are allowed.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Positive margin rate | 120 days
  Determine the positive margin status rate (based on the surgical pathology report) for the favorable cohort who successfully undergo reproductive organ sparing radical cystectomy

SECONDARY OUTCOMES:
Sexual function | 15 months
  Evaluate sexual function as measured by the Female Sexual Function Index (FSFI). The FSFI consists of 19 questions measuring female sexual function across six domains, including desire (2 items), arousal (4 items), lubrication (4 items), orgasm (3 items), satisfaction (3 items), and pain (3 items). Each response is assigned a score of either 0 to 5 or 1 to 5, with a higher score meaning a greater level of sexual functioning. The scores are summed to produce a composite score ranging from 4 to 36, with a higher score meaning better sexual functioning.
Quality of life | 15 months
  Evaluate quality of life as measured by the FACT-G questionnaire. The FACT-G measures various aspects of physical, social, emotional, and functional well-being over the past 7 days on a scale of 0-4 (with 0 meaning "Not at all" and 4 meaning "Very much").
Local recurrence | 12 months
  Determine the local recurrence rate.
Distant recurrence | 12 months
  Determine the distant recurrence rate.
Incidence rate of adjacent pelvic organ involvement | 12 months
  Determine the incidence of adjacent pelvic organ involvement in women undergoing radical cystectomy deemed "unfavorable" based on the decision tool.
Prediction of extravesicular disease | 15 months
  Evaluate the ability of staging MRI of the pelvis to predict extravesicular disease.
Prediction of adjacent pelvic organ involvement | 15 months
  Evaluate the ability of staging MRI of the pelvis to predict adjacent pelvic organ involvement

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Benidir, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States